CLINICAL TRIAL: NCT01071577
Title: Collection of Bone Marrow From Healthy Volunteers and Patients for the Production of Clinical Bone Marrow Stromal Cells (BMSC)Products
Brief Title: Collection of Bone Marrow From Healthy Volunteers and Patients for the Production of Clinical Bone Marrow Stromal Cell (BMSC) Products
Status: Terminated | Type: Observational
Why Stopped: The corresponding clinical trials have been completed or terminated; therefore, this study is no longer required to produce additional cells.
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 100053; 10-CC-0053
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Bone Marrow Stromal Cells
Keywords: Bone Marrow Stromal Cells; Mesenchymal Stem Cells; Immune Modulation; Tissue Regeneration; Natural History

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Healthy volunteers wanting to donate BMSC for allogeneic use
- Patients: Patients donating BMSC for autologous use

SUMMARY:
Background:

* Bone marrow stromal cells (BMSCs) can be grown from bone marrow provided by healthy volunteers. Volunteer bone marrow donors for BMSCs are generally required to meet the same healthy history and infectious disease marker screening criteria as volunteer blood donors. BMSCs are being used to treat a number of immune system and cardiovascular disorders, including graft-versus-host disease (GVHD), heart disease, and vascular disease. The National Institutes of Health Clinical Center is interested in collecting bone marrow aspirates and biopsies from healthy volunteers to produce clinical-grade BMSCs to treat Clinical Center patients.
* This study will also collect bone marrow from autologous donors (donors who will later receive their own BMSCs) for further treatment.

Objectives:

- To collect bone marrow aspirates and biopsies from healthy subjects and autologous donors in order to produce BMSCs.

Eligibility:

- Individuals at least 18 years of age who are either healthy volunteers or individuals who will need to receive their own BMSCs.

Design:

* Prospective healthy volunteers will be asked a series of questions designed to identify exposure to human immunodeficiency virus (HIV), hepatitis B or C, or other transfusion-transmitted diseases. A blood sample will be collected and tested for the abovementioned diseases and for other problems that may prevent bone marrow donation.
* Prospective autologous donors will also have blood tests to evaluate their own suitability for bone marrow donation.
* Eligible participants will be scheduled to provide a marrow aspirate/biopsy, taken from the upper part of the thigh bone, using standard bone marrow donation techniques.
* The collected bone marrow will be processed into BMSCs at the National Institutes of Health.

DETAILED DESCRIPTION:
Bone marrow stromal cells (BMSCs) can be grown from bone marrow aspirates and biopsies, and are being used to treat a number of disorders including: graft-versus-host disease (GVHD), ischemic heart disease, peripheral vascular disease and autoimmune diseases. The purpose of this protocol is to collect bone marrow aspirates and biopsies from healthy volunteers to produce clinical grade BMSCs to treat Clinical Center patients and to develop new methods for producing and assessing the quality of BMSCs. In some cases, the donors will be the recipients of the ex vivo expanded cells (autologous transplantation). In other cases, no matching of HLA or other antigens is required between the marrow donor and the BMSC recipient, so the donors will be required to meet the same healthy history and infectious disease marker screening criteria as volunteer blood donors. The BMSCs will be produced in the GMP Clinical Cell Processing Laboratory, located in the Cell Processing Section (CPS), Department of Transfusion Medicine (DTM), Clinical Center. After the BMSCs are produced by the Cell Processing Laboratory, they will be infused directly into Clinical Center patients on protocol, or cryopreserved and stored, and used as they are needed to treat Clinical Center patients. Up to 250 subjects will be enrolled in this study. This protocol will provide a mechanism for banking fresh and frozen BMSC products that can be used for patient care and research. This is not a treatment protocol. Subjects receiving these BMSC products will be enrolled in specific BMSC treatment protocols.

ELIGIBILITY:
* INCLUSION CRITERIA RELATED OR THIRD PARTY DONORS (ALLOGENEIC CELLS):
* Age greater than or equal to 18 years old
* Ability to give informed consent
* Adequate clinical parameters (all of the following):

  * Afebrile (temperature less than 38 (Infinite) C)
  * Systolic blood pressure greater than 100 & less than180 mmHg
  * Diastolic blood pressure greater than 50 & less than 100 mmHg
  * Heart rate between 40-100 beats/minute
* Females of child-bearing potential must have a negative pregnancy test and one of the following:

  * Be surgically sterile
  * Be abstinent until the marrow is collected
  * Use oral contraceptives, or other form of hormonal birth control
  * Use an intra-uterine device (IUD) as birth control
* Use (by ensuring her male partner(s) use(s) barrier contraception (condom) as birth control

INCLUSION CRITERIA AUTOLOGOUS DONORS

* Age greater than or equal to 18 years old
* Ability to give informed consent
* Females of child-bearing potential must have a negative pregnancy test and one of the following:

  * Be surgically sterile
  * Be abstinent until the marrow is collected
  * Use oral contraceptives, or other form of hormonal birth control
  * Use an intra-uterine device (IUD) as birth control
  * Use (by ensuring her male partner(s) uses) barrier contraception (condom) as birth control

EXCLUSION CRITERIA RELATED OR THIRD PARTY DONORS (ALLOGENEIC CELLS)

* Medical history that includes any of the following:

  * Thrombocytopenia or other blood dyscrasias
  * Bleeding diathesis
  * Antibiotic use within the prior 48 hours
  * History of cancer
  * History of exposure to transfusion transmitted diseases including HIV and hepatitis B and C as defined by the Standards for Blood Banking and Transfusion Services, American Association of Blood Banks.
  * Travel to an area where malaria is endemic as defined by the CDC (www.cdc.gov/travel).
  * At risk for the possible transmission of Creuzefeldt-Jackob Disease (CJD) and Variant Creuzefeldt-Jackob Disease (vCJD) as described in the FDA Guidance for Industry, January 9, 2002, Revised Preventive Measures to Reduce the Possible Risk of Transfusion of Creuzefeldt-Jackob Disease (CJD) and Variant Creuzefeldt-Jackob Disease (vCJD) by Blood and Blood Products
* If female, pregnant within the past 6 weeks
* Febrile (temperature greater than 38 (Infinite) C)
* Systolic blood pressure less than 100 or greater than 180 mmHg
* Diastolic blood pressure less than 50 or greater than 100 mmHg
* Heart rate less than 40 or greater than 100 beats/minute
* Anemia, thrombocytopenia, or leukopenia

  1. Hemoglobin level

     African American women < 11.5 grams/dL

     Other women < 12.0 grams/dL

     Men < 12.5 grams/dL
  2. HCT

     African American women < 34%

     Other women < 36%

     Men < 38%
  3. Platelets less than 150 x 10(3)/microL
  4. Absolute neutrophil count less than 1.0 x 10(3)/microL
* Prolonged coagulation assays

  1. PT greater than 15.2 seconds
  2. PTT greater than 37.3 seconds
* Positive tests for blood borne pathogens (as required by the Standards for Blood Banks and Transfusion Services, American Association of Blood Banks. The currently required tests include anti-HIV1/2, anti-HCV, Anti-HTVLI/II, anti-T. Cruzi, HBsAg, syphilis, and molecular testing for West Nile virus, HCV and HIV).
* Experiencing fever, malaise, anorexia, weight loss or night sweats consistent with active tuberculosis infection

EXCLUSION CRITERIA AUTOLOGOUS DONORS

-Medical history that includes any of the following:

* Currently Pregnant
* Positive tests for anti-HIV1/2, anti-HCV, or HBsAg
* Active tuberculosis infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers wanting to donate BMSC, may be NIH employees as well as Clinical Center patients.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2010-03-17 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-08-07 (Actual)

PRIMARY OUTCOMES:
Tissue Collection | At study visit
  Tissue Collection

CONTACTS AND LOCATIONS:
Overall Officials: David F Stroncek, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Jin P, Zhao Y, Liu H, Chen J, Ren J, Jin J, Bedognetti D, Liu S, Wang E, Marincola F, Stroncek D. Interferon-gamma and Tumor Necrosis Factor-alpha Polarize Bone Marrow Stromal Cells Uniformly to a Th1 Phenotype. Sci Rep. 2016 May 23;6:26345. doi: 10.1038/srep26345. PMID 27211104
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-CC-0053.html